CLINICAL TRIAL: NCT05994560
Title: Valor de la oclusión Temporal de Las Arterias Uterinas en la miomectomía Por Laparoscopia
Brief Title: The Value of Uterine Artery Occlusion in Laparoscopic Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, enrique moratalla bartolome, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 324/19
Record Dates: First submitted 2023-07-20; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Uterine Myomectomy
Keywords: myomectomy; temporary occlusion; uerine arteries

STUDY DESIGN:
Intervention Model Description: randomized clinical tria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without temporary occlusion (Other): Without temporary occlusion: No occlusion of uterine or útero-ovarian ligaments during laparoscopy myomectomy
  Interventions: Other: With temporary occlusion
- With temporary occlusion (Active Comparator): Temporary occlusion of the uterine arteries and utero-ovarian ligaments during laparoscopic myomectomy
  Interventions: Other: With temporary occlusion

INTERVENTIONS:
Other: With temporary occlusion — at the time of surgery the randomization table was consulted and if it was in the occlusion arm was performed

SUMMARY:
The objective of this study is to determine whether patients undergoing laparoscopic myomectomy with temporary occlusion of the uterine arteries and utero-ovarian ligaments using clips experience a decrease in blood loss during surgery compared to patients who undergo laparoscopic myomectomy without clips.

DETAILED DESCRIPTION:
Introduction:

Uterine fibroids are the most common benign tumors originating in the smooth muscle of the female genital tract. They occur in approximately 70% of women of middle age. Often, they cause abnormal uterine bleeding, pain, pelvic pressure, urinary and intestinal symptoms, and/or pregnancy complications. However, many fibroids are small and asymptomatic. About 25% of white women and 50% of black women will develop symptomatic fibroids. Fibroids are more common among overweight or obese women. Potential protective factors for fibroid occurrence are pregnancies and smoking, with a possible causal relationship, although the exact mechanism is not clear.

The treatment for women with uterine fibroids should be individualized based on their symptoms, size and location of fibroids, age, the need and desire to preserve fertility or the uterus, the availability of therapy, and the surgeon's experience. While hysterectomy is the definitive surgical treatment for symptomatic fibroids in women who do not wish to preserve fertility or their uterus, myomectomy is the treatment of choice for those with unfulfilled reproductive desires or a clear desire to keep their uterus and who are not suitable candidates for medical treatment.

The surgical planning for myomectomy should be based on the location, size, and number of fibroids, aided by appropriate imaging tests such as high-resolution ultrasound or magnetic resonance imaging (MRI).

Justification of the Study:

Intraoperative bleeding is one of the most frequent complications of laparoscopic myomectomy and may sometimes require transfusion. Therefore, methods that could reduce bleeding during surgery have been proposed, such as temporary occlusion of the uterine arteries and utero-ovarian ligaments. However, the efficacy and safety of this technique for use during laparoscopic myomectomy have not been clearly investigated.

Research Hypothesis:

The study aims to identify the efficacy of temporary occlusion of the uterine arteries during laparoscopic myomectomy.

Objectives:

Primary Objective:

- To compare the hemoglobin loss in g/dL (grams per deciliter) before and after surgery and intraoperative blood aspirate in milliliters between two groups of patients with symptomatic fibroids undergoing laparoscopic surgery, one with temporary occlusion of uterine arteries and utero-ovarian ligaments using clips and the other without such occlusion.

Secondary Objectives:

* To compare the surgical time of each technique.
* To compare the need for transfusion between both groups.
* To compare the improvement in symptoms for which the patients undergo surgery.
* To compare the length of hospital stay in each group.
* To compare possible complications of each technique.

Methodology:

Design:

A prospective randomized longitudinal study.

Study Subjects:

Patients with symptomatic fibroids requiring laparoscopic surgery as treatment, from the Gynecology Service of Hospital Ramón y Cajal and the HM Hospital, will be recruited. They will be randomized into two groups using simple random sampling. Patients will be given informed consent to participate in the study. The diagnosis of fibroids will be made through abdominal and/or transvaginal gynecological ultrasound and/or MRI.

Inclusion Criteria:

- Patients with uterine fibroids requiring surgical treatment via laparoscopy and with a desire to preserve the uterus.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.
* Women with symptomatic fibroids who are not candidates for laparoscopic surgery and/or have no desire to preserve the uterus.
* Patients for whom technical placement of clips during the intervention is not possible.

Main Variables:

* Preoperative and postoperative hemoglobin levels measured in g/dL.
* Intraoperative blood aspirate in milliliters.
* Surgical time.
* Need for transfusion.
* Improvement in symptoms.
* Length of hospital stay.
* Complications.

Data Collection:

The data will be collected from the patients' medical records and entered into a database using the SPSS software (version 23.0).

Ethical Aspects:

The study will follow the ethical principles laid out in the Declaration of Helsinki and Good Clinical Practice guidelines. Confidentiality of patient data will be maintained, and patients will provide informed consent to participate in the study.

Policy of Publications:

The study results will be published in scientific journals and medical conferences, subject to approval from the investigator and the Thesis Directors. The results will also be used as the basis for the investigator's doctoral thesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uterine fibroids requiring surgical treatment via laparoscopy and with a desire to preserve the uterus.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.
* Women with symptomatic fibroids who are not candidates for laparoscopic surgery and/or have no desire to preserve the uterus.
* Patients for whom technical placement of clips during the intervention is not possible.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Blood loss during surgery | during the time of the surgery
  The estimated intraoperative blood loss was calculated by measuring the amount of aspirated fluid at the end of the procedure minus the amount of fluid used for irrigation.

SECONDARY OUTCOMES:
To compare the surgical time of each technique | during surgery
  Time was recorded from the first skin incision to the last suture (minutes).
Length of hospital stay | until 1 week
  Days of hospital admission prior to discharge counting from the day of the intervention.
Difference in pre and postoperative hemoglobin levels (Hemoglobin loss) | up to 24 hours after surgery
  Preoperative hemoglobin was obtained within 24 hours before surgery, and postoperative hemoglobin was collected on postoperative day 1. Hemoglobin loss expressed in g/dL (grams per deciliter) was obtained from comparing hemoglobine pre and postoperative (before and after surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- Enrique Moratalla Bartolomé, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT05994560/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT05994560/ICF_001.pdf